CLINICAL TRIAL: NCT01472419
Title: Fluoropyrimidine/Platinum-based First-line Chemotherapy in Metastatic Esophageal Squamous Cell Carcinoma: Prognostic Factor Analysis in 239 Patients
Brief Title: Prognostic Factor Analysis in Metastatic Esophageal Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, Professor of Medicine, Sungkyunkwan University School of Medicine, Department of Hematology and Oncology, Samsung Medical Center
Other Study IDs: SMCESOPROGNOSIS
Record Dates: First submitted 2011-11-11; First posted 2011-11-16 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Metastatic Esophageal Squamous Cell Carcinoma
Keywords: metastatic esophageal squamous cell carcinoma; Fluoropyrimidine/platinum-based first-line chemotherapy; prognosis
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Esophageal squamous cell carcinoma is considerably more prevalent in East Asia. Despite of relatively high prevalence of esophageal SCC, prognosis is very poor with limited options of effective chemotherapy regimens. We attempted to identify favorable subgroups of patient who are likely to benefit from 5- fluorouracil/cisplatin(FP) or capecitabine/cisplatin (XP) chemotherapy as first-line treatment.Between January 2000 to December 2010, 239 patients were diagnosed of recurrent, metastatic esophageal SCC and received either FP or XP as first-line chemotherapy. Clinicopathologic variables and treatment outcome were retrospectively collected. we analysis treatment outcome of palliative chemotherapy in metastatic esophageal squamous cell carcinoma and make prognostic scoring system. The present study represents the largest series to analyze the treatment outcome of FP/XP chemotherapy in metastatic SCC. Risk-adapted stratification of treatment for subgroup of metastatic SCC patients should be actively pursued.

ELIGIBILITY:
Inclusion Criteria:

* recurrent, metastatic esophageal SCC
* received either FP or XP as first-line chemotherapy.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Between January 2000 to December 2010, 239 patients were diagnosed of recurrent, metastatic esophageal SCC and received either FP or XP as first-line chemotherapy.
Sampling Method: Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Jeeyun Lee, M.D., Ph.D., Principal Investigator — Samsung Medical Center, Seoul, Korea